CLINICAL TRIAL: NCT01897727
Title: Randomized Controlled Trial of Spironolactone Versus Standard of Care Blood Pressure Treatment on the Severity of Obstructive Sleep Apnea in Patients With Resistant Hypertension
Brief Title: Etiology of Sleep Apnea-related Hyperaldosteronism - BP Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Eric Judd, Sub investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F080821012; R01HL075614 (NIH)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2013-12

CONDITIONS: Obstructive Sleep Apnea; Resistant Hypertension; Hyperaldosteronism
Keywords: sleep apnea; hypertension; aldosterone; hyperaldosteronism; spironolactone; blood pressure; resistant
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hyperaldosteronism; Sleep Apnea Syndromes; Hypertension | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spironolactone (Active Comparator): Spironolactone 25 mg administered following baseline measurements and uptitrated to 50 mg if BP > 140/90 mm Hg throughout the 3 month study.
  Interventions: Drug: Spironolactone
- Standard of care BP treatment (Sham Comparator): Antihypertensive medication added and/or uptitrated to keep BP < 140/90 mm Hg throughout the study.
  Interventions: Drug: BP medication uptitration

INTERVENTIONS:
Drug: Spironolactone
  Arms: Spironolactone
Drug: BP medication uptitration — antihypertensive medication added or uptitrated following standard of care
  Arms: Standard of care BP treatment

SUMMARY:
Hypertension affects an estimated 60-70 million Americans, predisposing them to potentially life threatening cardiovascular complications. Resistant hypertension, defined as uncontrolled blood pressure on 3 or more different antihypertensive agents, is common, affecting 15-20% of the entire hypertensive population or an estimated 12-14 million Americans. Although associated with obesity, increasing age, black race, and chronic kidney disease, mechanisms of treatment resistance remain obscure. The investigators' laboratory identified primary aldosteronism (PA) as a common cause of treatment resistance with a prevalence of 20% among subjects with resistant hypertension. This is clinically important because recognition of PA can lead to effective treatment with use of aldosterone blockers. Obstructive sleep apnea (OSA) is strongly associated with and predicts development of hypertension as demonstrated in landmark cohort studies including the Sleep Heart Health Study and the Wisconsin Sleep Cohort Study.

The investigators' laboratory has confirmed OSA to be extremely common in subjects with resistant hypertension, with a prevalence of approximately 85%. Recognizing that PA and OSA are exceptionally common in subjects with resistant hypertension, the investigators hypothesized that the 2 may be causally related. In testing this hypothesis, the investigators recently reported that plasma aldosterone levels are positively correlated with OSA severity in subjects with resistant hypertension but not in normotensive control subjects. This observation suggests that there is an important mechanistic interaction between untreated OSA and aldosterone excess in subjects with resistant hypertension. While the investigators' original hypothesis was that OSA stimulates aldosterone release, the investigators recognize that the opposite may also be true; that is, aldosterone excess in subjects with resistant hypertension worsens OSA. Distinguishing between these two possibilities has potentially far-reaching clinical implications. If the former hypothesis is true, effective treatment of OSA would be expected to suppress aldosterone release in subjects with resistant hypertension, thereby reversing the underlying cause of their treatment resistance. If the latter hypothesis is true, use of mineralocorticoid receptor antagonists would be expected to reduce OSA severity in subjects with resistant hypertension, thereby enhancing treatment of OSA. Either scenario would represent a new treatment approach for a highly prevalent and serious medical problem.

ELIGIBILITY:
Inclusion Criteria:

* Resistant hypertension defined as office BP that is uncontrolled with 3 or more antihypertensive medications
* Moderate-severe OSA defined as AHI ≥15 events/hr
* Self-reported adherence >80% with prescribed antihypertensive medications.

Exclusion Criteria:

* Ongoing use of a potassium sparing diuretic
* History of congestive heart failure (ejection fraction of <40%)
* Chronic kidney disease (creatinine clearance <60 ml/min)
* History of cardiovascular disease (stroke, TIA, myocardial infarction, or revascularization procedure)
* Known or suspected history of secondary cause of hypertension other than primary aldosteronism
* Severe nocturnal hypoxemia (O2 desaturation nadir <60%)
* White coat hypertension defined as office BP >140/90 mm Hg and ambulatory daytime BP <135/85 mm Hg
* Central sleep apnea (defined as 5% or more of the apneas as central apneas) and/or the presence of any Cheyne-Stokes breathing
* Subjects working shift work or having other known circadian rhythm disorders such that their sleep-wake schedule is altered
* Excessive daytime sleepiness as indicated by an Epworth score of >10
* Pregnant Women

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-01; Primary Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Gaddam K, Pimenta E, Thomas SJ, Cofield SS, Oparil S, Harding SM, Calhoun DA. Spironolactone reduces severity of obstructive sleep apnoea in patients with resistant hypertension: a preliminary report. J Hum Hypertens. 2010 Aug;24(8):532-7. doi: 10.1038/jhh.2009.96. Epub 2009 Dec 17. PMID 20016520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive adult patients with symptoms of OSA and resistant HTN between 2009 to 2012, were enrolled from the Hypertension Clinic at the University of Alabama at Birmingham.
Pre-assignment Details: There was no wash out; ongoing use of a potassium sparing diuretic, including spironolactone, eplerenone, triamterene, or amiloride precluded study participation.
  A total of 17 participants (out of the 41 who were enrolled) were randomized into the two groups. 24 participants met exclusion criteria before randomization.
Period: Overall Study
Arm/Group | Spironolactone | Standard of Care BP Treatment
Started | 8 | 9
Completed | 8 | 8
Not Completed | 0 | 1
Not completed — Exclusion: central sleep apnea | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spironolactone | Standard of Care BP Treatment | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (8.3) | 56.8 (6.3) | 58.4 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Severity of Obstructive Sleep Apnea
Description: 3 month change in apnea-hypopnea index assessed by diagnostic, full-night polysomnography. AHI values are typically categorized as 5-15/hr = mild; 15-30/hr = moderate; and > 30/h = severe.
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Spironolactone | Standard of Care BP Treatment
Number analyzed (Participants) | 8 | 8
events/hour | -18.3 (16.1) | 7.0 (30.0)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Spironolactone | Standard of Care BP Treatment
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
1. Unanticipated enrollment challenges led to small numbers of participants analyzed.
2. Open-label study design may have prevented a placebo effect.
3. An outlier in AHI was present in the control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes